CLINICAL TRIAL: NCT01096342
Title: Phase II Trial of Cdk Inhibitor SCH 727965 in Multiple Myeloma
Brief Title: Dinaciclib in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02795; NCI-2012-02795 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MAYO-MC0888; MC0888 (Other: Mayo Clinic); 8288 (Other: CTEP); P30CA015083 (NIH); N01CM62205 (NIH)
Record Dates: First submitted 2010-03-30; First posted 2010-03-31 (Estimated); Results first posted 2013-02-25 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2013-12

CONDITIONS: Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — dinaciclib

ARMS (1):
- Treatment (Experimental): Patients receive dinaciclib IV over 2 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: dinaciclib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: dinaciclib — Given IV
  Other Names: CDK inhibitor SCH 727965; cyclin-dependent kinase inhibitor SCH 727965; SCH 727965
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well giving dinaciclib works in treating patients with relapsed or refractory multiple myeloma. Dinaciclib may stop the growth of cancer cells by clocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy (overall response rate) of single agent SCH 727965 in patients with relapsed or refractory multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the toxicities associated with use of single agent SCH 727965 in patients with relapsed or refractory multiple myeloma.

II. To evaluate the response duration and progression free survival among patients with relapsed or refractory multiple myeloma undergoing treatment with single agent SCH 727965.

III. To study the effect of SCH 727965 on myeloma cell proliferation, apoptotic rates and to assess the ability of the drug to inhibit drug targets (cyclin dependent kinases, cdk in the myeloma cell.

OUTLINE: This is a multicenter, dose-escalation study.

Patients receive dinaciclib IV over 2 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Blood and bone marrow samples are collected periodically for correlative studies. (US sites only)

After completion of study treatment, patients are followed up for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory multiple myeloma
* Measurable disease as defined by at least ONE of the following:

  * Serum monoclonal protein >= 1.0 g/dL
  * > 200 mg of monoclonal protein in the urine on 24 hour electrophoresis
  * Serum immunoglobulin free light chain >= 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
* ≤ 5 prior therapies; stem cell transplantation and preceding induction therapy will be considered as one therapy; NOTE: Patients must not be candidates for stem cell transplantation or should have had stem cells collected previously
* Life expectancy of ≥ 3 months
* ECOG performance status of 0, 1 or 2
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 75,000/mcL
* Hemoglobin >= 8 g/dL
* Total serum bilirubin within normal institutional limits
* AST (SGOT)/ALT(SGPT) =< 2.5 X institutional ULN
* Creatinine < 2.5 mg/dL
* Negative serum pregnancy test done ≤7 days prior to registration (for women of childbearing potential only); NOTE: Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* Willingness to provide blood and bone marrow samples for mandatory research component of this study; (US sites only)

Exclusion Criteria:

* Any of the following prior therapies:

  * Myelosuppressive therapy for myeloma ≤ 3 weeks prior to registration or those who have not recovered from acute reversible adverse events due to agents administered > 3 weeks earlier
  * Non-myelosuppressive agents like thalidomide or high dose corticosteroids ≤ 2 weeks prior to registration
* Receiving any other investigational agents
* Concomitant high dose corticosteroids

  * NOTE: Concurrent use of corticosteroids, but patients may be on chronic steroids (maximum dose 20 mg/day prednisone equivalent) if they are being given for disorders other than amyloid, i.e., adrenal insufficiency, rheumatoid arthritis, etc.
  * NOTE: Bisphosphonates are considered to be supportive care rather than therapy, and are thus allowed while on protocol treatment
* Active malignancy with the exception of non melanoma skin cancer or in situ cervical or breast cancer
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infections or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or nursing women; NOTE: Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with SCH 727965, breastfeeding should be discontinued if the mother is treated with SCH 727965
* Currently taking inhibitors/inducers of CYP3A4; (SCH 727965 metabolizes via the CYP3A4 enzyme; there are potential drug interactions with concomitant use of CYP3A4 potent inhibitors/inducers; Principal Investigator should review each case and determine if patients on the CYP3A4 potent inhibitors/inducers are eligible and will make all effort to switch to alternative drugs; patients should not take grapefruit/ grapefruit juice or St. Johns' Wort)
* Men or women of childbearing potential who are unwilling to employ adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-07; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaji Kumar, Principal Investigator — Mayo Clinic
Locations (6):
- United States (5):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Kumar SK, LaPlant B, Chng WJ, Zonder J, Callander N, Fonseca R, Fruth B, Roy V, Erlichman C, Stewart AK; Mayo Phase 2 Consortium. Dinaciclib, a novel CDK inhibitor, demonstrates encouraging single-agent activity in patients with relapsed multiple myeloma. Blood. 2015 Jan 15;125(3):443-8. doi: 10.1182/blood-2014-05-573741. Epub 2014 Nov 13. PMID 25395429

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 7/2009 to 12/2011, 29 participants were accrued. The study opened at 50 mg/m^2, accrued 2, and closed for safety review and protocol amendment. The study reopened with a dose escalation phase and accrued 4 at 30 mg/m^2 dose, 7 at 40 mg/m^2 dose, and 6 at 50 mg/m^2 dose. The Phase II dose level was set at 50 mg/m^2 and accrued 10 participants.
Pre-assignment Details: Of the 10 participants accrued in the Phase II portion of the study, one was excluded for protocol violation. The 6 participants treated in the Safety Analysis Phase at the 50 mg/m^2 dose level (after the protocol amendment) are included in the Phase II analysis. Therefore, this Phase II analysis is based on 15 evaluable participants.
Groups:
- Phase II: 50 mg/m^2: Participants were accrued at 50 mg/m^2 dose level after December 30, 2009 addendum. Participants to receive 50 mg/m^2 dinaciclib IV over 2 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Phase II: 50 mg/m^2
Started | 16
Completed | 15
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: A total of sixteen participants were accrued to the 50 mg/m^2 after the December 30, 2009 amendment (6 at MTD plus 10 phase II) and were grouped together as Phase II. Of these 16 particpants, one participant was excluded due to a major treatment violation.
Groups:
- Phase II: Participants were accrued at 50 mg/m^2 dose level after December 30, 2009 addendum. Participants to receive 50 mg/m^2 dinaciclib IV over 2 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Phase II
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 64 [55 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 12
  Singapore | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Confirmed Responses, Defined to be an sCR, CR, VGPR, or PR Noted as the Objective Status on Two Consecutive Evaluations.
Description: Complete Response (CR):
  Negative immunofixation of serum and urine Normalization of FLC ratio < 5% plasma cells in bone marrow Disappearance of any soft tissue plasmacytomas
  Stringent Complete Response (sCR):
  CR, as above, with absence of clonal cells in bone marrow
  Partial Response (PR):
  One of the following:
  1. A ≥ 50% reduction of measurable serum M-protein.
  2. A reduction in 24h measurable urinary M-protein by ≥ 90% or to <200 mg per 24h.
  3. A ≥ 50% decrease in the difference between involved and uninvolved FLC levels.
  4. ≥50% reduction in bone marrow plasma cells is required in place of Mprotein, provided baseline percentage was ≥ 30%
  5. A ≥50% reduction in the size of soft tissue plasmacytomas.
  Very Good Partial Response (VGPR):
  PR as defined above in addition to having serum and urine M-component detectable by immunofixation but not on electrophoresis.
Time Frame: Up to 3 years
Population: Fifteen of the 16 accrued Phase II participants were analyzed (1 participant was a protocol violation).
Measure: Number; unit: participants
Arm/Group | Phase II
Number analyzed (Participants) | 15
participants
  Complete Response (CR) | 0
  Stringent Complete Response (sCR) | 0
  Very Good Partial Response (VGPR) | 0
  Partial Response (PR) | 0

2. Secondary Outcome: Progression-free Survival
Description: The distribution of progression-free survival will be estimated using the method of Kaplan-Meier.
Time Frame: Time from registration to progression or death due to any cause, assessed up to 3 years
Population: All 15 evaluable participants were analyzed for Progression-Free Survival.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II
Number analyzed (Participants) | 15
months | 2.73 [0.69 to 5.52]

3. Secondary Outcome: Duration of Response
Description: The distribution of duration of response will be estimated using the method of Kaplan-Meier.
Time Frame: Date at which the patient's objective status is first noted to be either an sCR, CR, PR, or VGPR to the earliest date progression is documented, assessed up to 3 years
Population: Duration of Response was not analyzed due to lack of responses.
Arm/Group | Phase II
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Phase II: 50 mg/m^2
Serious Adverse Events (participants affected / at risk) | 7/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase II: 50 mg/m^2 (N=15)
Dry eye syndrome (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Leukocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase II: 50 mg/m^2 (N=15)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (3)
Vision blurred (Eye disorders) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 12 (28)
Nausea (Gastrointestinal disorders) | 9 (19)
Vomiting (Gastrointestinal disorders) | 6 (8)
Fatigue (General disorders) | 14 (27)
Fever (General disorders) | 3 (3)
Pain (General disorders) | 1 (2)
Peripheral nerve infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (2)
Alanine aminotransferase increased (Investigations) | 5 (8)
Aspartate aminotransferase increased (Investigations) | 7 (18)
Bilirubin increased (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 6 (9)
Lymphocyte count decreased (Investigations) | 5 (10)
Neutrophil count decreased (Investigations) | 4 (5)
Platelet count decreased (Investigations) | 11 (19)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (3)
Peripheral motor neuropathy (Nervous system disorders) | 2 (11)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (19)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (6)
Hypotension (Vascular disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less